CLINICAL TRIAL: NCT07049900
Title: Baby ABS (Abdominal Binder Study) : Impact of Abdominal Binder Use on Abdominal Wall Development in Premature Infants Requiring CPAP Support
Brief Title: Baby ABS (Abdominal Binder Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PEDS-2025-33787
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Premature; Premature Lungs; Ventilator Lung; Newborn; Rectus Abdominis
Keywords: bCPAP; CPAP; NAVA CPAP
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NeoBelllyBand (Active Comparator): Infants in this group will continue to have standard NICU care, with the addition of wearing the NeoBellyBand device while they remain on CPAP.
  Interventions: Device: NeoBelly Band
- Standard NICU Care (No Intervention): Infants in this group will receive standard neonatal intensive unit care as defined by the University of Minnesota Masonic Children's Hospital NICU protocol.

INTERVENTIONS:
Device: NeoBelly Band — The DandleLion NeoBellyBand (NBB) is an FDA listed Class 1 medical device that is 510k exempt and is categorized under therapeutic medical binders. This device is indicated to be used while the infant is receiving CPAP support in order to reduce CBS. The NBB is made of a medical-grade blend of fabric and foam that is latex and neoprene-free and is reported as safe to use on premature infant skin. There are two sizes available and the outer fabric is attached with adjustable Velcro. It is a single baby use and may be hand washed and reused. This device is currently in use in multiple NICUs around the country, and as it has already been FDA-approved for the purpose of our investigation.
  Arms: NeoBelllyBand

SUMMARY:
The primary outcome of this study is to determine if the use of the FDA-approved DandleLion NeoBellyBand increases the thickness of the rectus abdominis muscle in premature babies receiving continuous positive pressure ventilation, leading to infants reaching full oral feedings at an earlier corrected gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Premature viable neonates with corrected gestational age of 26-31 weeks
* Anticipated to require non-invasive continuous positive pressure ventilation including bCPAP, CPAP, and NAVA CPAP for a minimum of 2 weeks either on their first trial of CPAP or after extubation.

Exclusion Criteria:

* Outside of gestational age at birth
* Umbilical lines
* Genetic condition or neuromuscular anomaly
* Known abdominal anomaly
* Non-viable neonates and neonates with uncertain viability who are not anticipated to be able to survive with standard NICU care.
* Surgical intervention on the abdominal wall, such as gastroschisis or history of surgical NEC
* Compromised skin integrity of abdominal wall
* Any condition in the opinion of the investigator that would risk the data integrity or collection of the study

Ages: 26 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in thickness of the rectus abdominis muscle | 8 weeks
  Thickness measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ramel, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No